CLINICAL TRIAL: NCT03630952
Title: A Multicenter, Double-Masked, Randomized, Dose-Ranging Trial to Evaluate the Efficacy and Safety of Conbercept Intravitreal Injection in Subjects With Neovascular Age-Related Macular Degeneration (AMD) (PANDA-2)
Brief Title: Efficacy and Safety Trial of Conbercept Intravitreal Injection for Neovascular AMD (PANDA-2)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: desired primary endpoint was not met
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHB-1802
Record Dates: First submitted 2018-08-11; First posted 2018-08-15 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — KH902 fusion protein; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 mg Conbercept (Experimental): Subjects received 0.5 mg conbercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every eight weeks thereafter (0.5 mg, q8w) through Week 36. At the Week 40 visit, the criteria-based pro re nata (PRN) approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Interventions: Biological: 0.5 mg Conbercept Intravitreal Injection
- 1.0 mg Conbercept (Experimental): Subjects received 1.0 mg conbercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every twelve weeks thereafter (1.0 mg, q12w) through Week 36. At the Week 40 visit, the criteria-based PRN approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Interventions: Biological: 1.0 mg Conbercept Intravitreal Injection
- Aflibercept (Active Comparator): Subjects received 2.0 mg aflibercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every eight weeks thereafter (2.0 mg, q8w) through Week 36. At the Week 40 visit, the criteria-based PRN approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Interventions: Biological: 2.0 mg Aflibercept Intravitreal Injection

INTERVENTIONS:
Biological: 0.5 mg Conbercept Intravitreal Injection — Subjects received 0.5 mg conbercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every eight weeks thereafter (0.5 mg, q8w) through Week 36. At the Week 40 visit, the criteria-based pro re nata (PRN) approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Arms: 0.5 mg Conbercept
Biological: 1.0 mg Conbercept Intravitreal Injection — Subjects received 1.0 mg conbercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every twelve weeks thereafter (1.0 mg, q12w) through Week 36. At the Week 40 visit, the criteria-based PRN approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Arms: 1.0 mg Conbercept
Biological: 2.0 mg Aflibercept Intravitreal Injection — Subjects received 2.0 mg aflibercept intravitreal injection at Day 1, Week 4 and Week 8 (three injection loading dose), and treated every eight weeks thereafter (2.0 mg, q8w) through Week 36. At the Week 40 visit, the criteria-based PRN approach will begin through the end of the treatment period at Week 92, for a total of 92 weeks treatment in the study eye.
  Other Names: Eylea®
  Arms: Aflibercept

SUMMARY:
The purpose of this clinical study is to evaluate the efficacy and safety of two different levels of conbercept intravitreal (IVT) injection as compared to the approved vascular endothelial growth factor (VEGF) antagonist active control, aflibercept intravitreal injection (2.0 mg/eye, Eylea®), in subjects with neovascular AMD.

DETAILED DESCRIPTION:
A multicenter, multinational, double-masked, parallel-group, dose-ranging, active-controlled, randomized trial, which will randomize approximately 1140 subjects in a ratio of 1:1:1 to receive IVT injections of 0.5 mg conbercept, 1.0 mg conbercept, or 2.0 mg aflibercept. The trial includes a screening period of less than or equal to 14 days, followed by a treatment period of 92 weeks (last assessment at 96 weeks) with primary efficacy analysis at 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 50 years of age at the Screening visit;
2. Females must be at least 1 year postmenopausal, or surgically sterilized, or, if of childbearing potential, must have a negative pregnancy test at the Screening visit;

   o Women of childbearing potential must agree to use a highly effective method of contraception throughout the study.
3. Have received no previous treatment for neovascular AMD, including laser photocoagulation and/or photodynamic therapy (PDT) and/or IVT VEGF antagonists (treatment naïve) and;
4. Have active subfoveal choroidal neovascularization (CNV) lesions secondary to AMD (including polypoidal choroidal vasculopathy (PCV)) evidenced by subfoveal fluorescein angiography (FA) leakage, or definite subfoveal fluid by SD-OCT in the study eye at Screening;
5. Have a ETDRS BCVA letter score of 78 to 25 in the study eye at Screening;
6. Are willing and able to sign the study written informed consent form (ICF).

Exclusion Criteria:

1. Have had any prior ocular or systemic treatment (investigational or approved) or surgery for the treatment of neovascular AMD in the study eye except dietary supplements or vitamins;
2. Have participated as a subject in any interventional clinical trial within one month (30 days) prior to Baseline visit;
3. Have a subretinal hemorrhage that is either 50% or more of the total lesion area, or blood is under the fovea and is one or more disc areas in size (greater than 2.5 mm2) in the study eye at Screening;
4. Have any retinal pigment epithelial tears or rips in the study eye at Screening or upon examination at Baseline;
5. Have any vitreous hemorrhage in the study eye upon examination at Baseline or history of vitreous hemorrhage within eight weeks prior to Screening;
6. Have any other cause of CNV;
7. Have had prior pars plana vitrectomy in the study eye;
8. Have presence of a full thickness macular hole at Screening or upon examination at Baseline or a history of a full thickness macular hole in the study eye;
9. Have prior trabeculectomy or other filtration surgery in the study eye;
10. Have uncontrolled glaucoma;
11. Have active intraocular inflammation in either eye at Screening or upon examination at Baseline or a history of uveitis in either eye;
12. Have aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of yttrium aluminum garnet (YAG) posterior capsulotomy) in the study eye.
13. Significant media opacities, including cataract, in the study eye that, in the opinion of the Investigator, could require either medical or surgical intervention during the study period;
14. Have any use of long acting intraocular steroids, including implants, within six months prior to Day 1, Baseline;
15. Have any known allergy to povidone iodine or known serious allergy to the fluorescein sodium for injection in angiography;
16. Any history of known contraindications indicated in the Food and Drug Administration (FDA)-approved label for the active control;
17. If female, be pregnant (positive urine pregnancy test at Screening) or breastfeeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in best corrected visual acuity (BCVA) at Week 36 in the study eye | Baseline to Week 36
  BCVA was assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) method

SECONDARY OUTCOMES:
Proportion of subjects maintaining vision (i.e., losing <15 ETDRS BCVA letters) from baseline to Week 36 | Baseline to Week 36
  To Assess Proportion of subjects maintaining vision (i.e., losing <15 ETDRS BCVA letters) from baseline to Week 36
Proportion of subjects gaining ≥15 ETDRS BCVA letters from baseline to Week 36 | Baseline to Week 36
  To Assess Proportion of subjects gaining ≥15 ETDRS BCVA letters from baseline to Week 36
Mean change from baseline in central retinal thickness (µm) by spectral domain optical coherence tomography (SD-OCT) at Week | Baseline and Week 36
  To Assess Mean change from baseline in central retinal thickness (µm) by spectral domain optical coherence tomography (SD-OCT) at Week
Proportion of subjects maintaining vision (i.e. losing <15 ETDRS BCVA letters) from baseline to Week 48 | Baseline to Week 48
  To Assess Proportion of subjects maintaining vision (i.e. losing <15 ETDRS BCVA letters) from baseline to Week 48
Mean change from baseline in ETDRS BCVA letter score at Week 96 | Baseline and Week 96
  To Assess Mean change from baseline in ETDRS BCVA letter score at Week 96
Number of participants with adverse events as measure of safety and tolerability | Baseline to Week 96
  To Assess Number of participants with adverse events as measure of safety and tolerability
Blood concentration of conbercept doses conducted in a subgroup of subjects, when feasible | Baseline to Week 96
  To Assess Blood concentration of conbercept doses conducted in a subgroup of subjects, when feasible
Half-life (t1/2) of conbercept doses conducted in a subgroup of subjects, when feasible | Baseline to Week 96
  To Assess Half-life (t1/2) of conbercept doses conducted in a subgroup of subjects, when feasible
Presence of anti-drug antibody of conbercept doses conducted in a subgroup of subjects, when feasible | Baseline to Week 96
  To Assess Presence of anti-drug antibody of conbercept doses conducted in a subgroup of subjects, when feasible

CONTACTS AND LOCATIONS:
Overall Officials: Yan Cheng, MD, PhD, Study Director — Chengdu Kanghong Biotechnology Co.,Ltd.
Locations (125):
- United States (64):
  - Kanghong Investigative Site, Phoenix, Arizona
  - Kanghong Investigative Site, Springdale, Arkansas
  - Kanghong Investigative Site, Arcadia, California
  - Kanghong Investigative Site, Bakersfield, California
  - Kanghong Investigative Site, Encino, California
  - Kanghong Investigative Site, Glendale, California
  - Kanghong Investigative Site, Glendora, California
  - Kanghong Investigative Site, Huntington Beach, California
  - Kanghong Investigative Site, Pasadena, California
  - Kanghong Investigative Site, Poway, California
  - Kanghong Investigative Site, Redlands, California
  - Kanghong Investigative Site, Riverside, California
  - Kanghong Investigative Site, San Francisco, California
  - Kanghong Investigative Site, Santa Barbara, California
  - Kanghong Investigative Site, Colorado Springs, Colorado
  - Kanghong Investigative Site, Waterford, Connecticut
  - Kanghong Investigative Site, Boynton Beach, Florida
  - Kanghong Investigative Site, Bradenton, Florida
  - Kanghong Investigative Site, Miami, Florida
  - Kanghong Investigative Site, Stuart, Florida
  - Kanghong Investigative Site, Winter Haven, Florida
  - Kanghong Investigative Site, Atlanta, Georgia
  - Kanghong Investigative Site, Augusta, Georgia
  - Kanghong Investigative Site, Marietta, Georgia
  - Kanghong Investigative Site, Elmhurst, Illinois
  - Kanghong Investigative Site, Indianapolis, Indiana
  - Kanghong Investigative Site, New Albany, Indiana
  - Kanghong Investigative Site, Leawood, Kansas
  - Kanghong Investigative Site, Springfield, Massachusetts
  - Kanghong Investigative Site, Grand Rapids, Michigan
  - Kanghong Investigative Site, Traverse City, Michigan
  - Kanghong Investigative Site, St Louis, Missouri
  - Kanghong Investigative Site, Reno, Nevada
  - Kanghong Investigative Site, Northfield, New Jersey
  - Kanghong Investigative Site, Teaneck, New Jersey
  - Kanghong Investigative Site, Albuquerque, New Mexico
  - Kanghong Investigative Site, Brooklyn, New York
  - Kanghong Investigative Site, Great Neck, New York
  - Kanghong Investigative Site, Liverpool, New York
  - Kanghong Investigative Site, Shirley, New York
  - Kanghong Investigative Site, Asheville, North Carolina
  - Kanghong Investigative Site, Winston-Salem, North Carolina
  - Kanghong Investigative Site, Youngstown, Ohio
  - Kanghong Investigative Site, Oklahoma City, Oklahoma
  - Kanghong Investigative Site, Medford, Oregon
  - Kanghong Investigative Site, Portland, Oregon
  - Kanghong Investigative Site, Springfield, Oregon
  - Kanghong Investigative Site, Camp Hill, Pennsylvania
  - Kanghong Investigative Site, Kingston, Pennsylvania
  - Kanghong Investigative Site, Ladson, South Carolina
  - Kanghong Investigative Site, Rapid City, South Dakota
  - Kanghong Investigative Site, Arlington, Texas
  - Kanghong Investigative Site, Austin, Texas
  - Kanghong Investigative Site, Bellaire, Texas
  - Kanghong Investigative Site, Dallas, Texas
  - Kanghong Investigative Site, Fort Worth, Texas
  - Kanghong Investigative Site, Kingwood, Texas
  - Kanghong Investigative Site, McAllen, Texas
  - Kanghong Investigative Site, Midland, Texas
  - Kanghong Investigative Site, Temple, Texas
  - Kanghong Investigative Site, Salt Lake City, Utah
  - Kanghong Investigative Site, Burlington, Vermont
  - Kanghong Investigative Site, Charlottesville, Virginia
  - Kanghong Investigative Site, Bellevue, Washington
- Bulgaria (3):
  - Kanghong Investigative Site, Plovdiv
  - Kanghong Investigative Site, Sofia
  - Kanghong Investigative Site, Varna
- China (3):
  - Kanghong Investigative Site, Beijing, Beijing Municipality
  - Kanghong Investigative Site, Shanghai, Shanghai Municipality
  - Kanghong Investigative Site, Tianjin, Tianjin Municipality
- Czechia (2):
  - Kanghong Investigative Site, Brno
  - Kanghong Investigative Site, Prague
- Denmark (5):
  - Kanghong Investigative Site, Aalborg
  - Kanghong Investigative Site, Aarhus N
  - Kanghong Investigative Site, Glostrup Municipality
  - Kanghong Investigative Site, Roskilde
  - Kanghong Investigative Site, Sønderborg
- France (8):
  - Kanghong Investigative Site, Bordeaux
  - Kanghong Investigative Site, Créteil
  - Kanghong Investigative Site, Dijon
  - Kanghong Investigative Site, Marseille
  - Kanghong Investigative Site, Paris
  - Kanghong Investigative Site, Poitiers
  - Kanghong Investigative Site, Saint-Cyr-sur-Loire
  - Kanghong Investigative Site, Strasbourg
- Hungary (5):
  - Kanghong Investigative Site, Pécs, Baranya
  - Kanghong Investigative Site, Szeged, Csongrád megye
  - Kanghong Investigative Site, Debrecen, Hajdú-Bihar
  - Kanghong Investigative Site, Budapest, Pest County
  - Kanghong Investigative Site, Zalaegerszeg, Zala County
- Israel (10):
  - Kanghong Investigative Site, Ashkelon, Ha'Darom
  - Kanghong Investigative Site, Beersheba
  - Kanghong Investigative Site, Haifa
  - Kanghong Investigative Site, Jerusalem
  - Kanghong Investigative Site, Kfar Saba
  - Kanghong Investigative Site, Petah Tikva
  - Kanghong Investigative Site, Poria – Neve Oved
  - Kanghong Investigative Site, Rehovot
  - Kanghong Investigative Site, Tel Aviv
  - Kanghong Investigative Site, Zrifin
- Italy (7):
  - Kanghong Investigative Site, Chieti
  - Kanghong Investigative Site, Florence
  - Kanghong Investigative Site, Genova
  - Kanghong Investigative Site, Milan
  - Kanghong Investigative Site, Negrar
  - Kanghong Investigative Site, Roma
  - Kanghong Investigative Site, Udine
- Kanghong Investigative Site, Riga, Latvia
- Slovakia (3):
  - Kanghong Investigative Site, Bratislava
  - Kanghong Investigative Site, Trenčín
  - Kanghong Investigative Site, Žilina
- United Kingdom (14):
  - Kanghong Investigative Site, Westcliff-on-Sea, Essex
  - Kanghong Investigative Site, Southampton, Hampshire
  - Kanghong Investigative Site, Gorleston-on-Sea, Norfolk
  - Kanghong Investigative Site, Frimley, Surrey
  - Kanghong Investigative Site, Belfast
  - Kanghong Investigative Site, Bradford
  - Kanghong Investigative Site, Bristol
  - Kanghong Investigative Site, Canterbury
  - Kanghong Investigative Site, Derby
  - Kanghong Investigative Site, Gorleston-on-Sea
  - Kanghong Investigative Site, Leeds
  - Kanghong Investigative Site, London
  - Kanghong Investigative Site, Sheffield
  - Kanghong Investigative Site, Sunderland

IPD SHARING:
Plan to Share IPD: No